CLINICAL TRIAL: NCT01530672
Title: Evaluation of the MBio Combined Syphilis/HIV Point-of-Care Diagnostic Test
Acronym: MBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS647
Record Dates: First submitted 2012-01-23; First posted 2012-02-10 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: HIV; Syphilis
Keywords: HIV; Syphilis; Combination; POC; point-of-care; MBIO
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ANC clients (Experimental)
  Interventions: Device: MBIO POC combined HIV syphilis test ( SnapEsi)

INTERVENTIONS:
Device: MBIO POC combined HIV syphilis test ( SnapEsi) — Venipuncture for routine ANC screening plus additional for device validation purposes.
  Other Names: MBIO; SnapEsi-beta HIV-1/Syphilis

SUMMARY:
This is a diagnostic validation study for a combined Syphilis/HIV test made by MBio Diagnostics, Inc (MBio, Boulder, CO, USA). Although the MBio Syphilis/HIV diagnostic platform is designed for use at point of care (POC), it is made to provide similar performance as reference standards. Diagnosing HIV and syphilis accurately with a single POC test will save time for clinic health workers and technicians, reduce loss-to follow-up caused by lengthy delays for lab-based tests, and save costs by eliminating the need for multiple tests. For this study, the sensitivity and specificity of the MBio HIV/Syphilis Serology System point-of-care diagnostic test will be determined using reference tests performed under controlled laboratory conditions. For this, clients receiving routine care in the ANCs at the New Nyanza Provincial General Hospital (NNPGH) and Kisumu District Hospital (KDH) will be consented to provide blood for the proposed study. Study volunteers will receive HIV and syphilis rapid tests provided as part of routine care, and will donate an additional blood for evaluating the MBio test against the reference tests in a laboratory setting. This study is an investigational prototype, not for product registration. The results from this study will be used to inform product development of a second iteration of the MBio device design. At the time that the device is ready to be registered, it will undergo another field evaluation at which time it will be submitted to the appropriate regulatory body. Because the MBIO device is an HIV test, the device would be submitted to National AIDS & STI Control Program (NASCOP), which is the appropriate regulatory body for HIV tests in Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Attending her first routine ANC visit and willing to undergo tests for HIV/syphilis
* Able and willing to legally consent for enrollment
* Able to demonstrate-comprehension of study details as they are explained in the consent process by passing all the test questions of understanding. The subject is only allowed two attempts at passing the test of understanding.

Exclusion Criteria:

* Unwilling to provide written informed consent.
* Unable to legally consent (minor without guardian)
* Opt out of HIV or syphilis test
* Previously diagnosed with autoimmune disorder (lupus, Lyme disease), as determined by client recollection or clinical record.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2900 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Device sensitivity/specificity | same-day
  Sensitivity & specificity of the MBIO device against HIV and syphilis reference tests

SECONDARY OUTCOMES:
Percent agreement with clinical diagnosis | same-day
  Percent agreement with HIV & syphilis rapid tests completed at clinic

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Steele, Ph.D, M.P.H., Principal Investigator — PATH; John Waitumbi, Ph.D, D.V.M., Principal Investigator — Walter Reed Project; Kathleen Tietje, PhD, Principal Investigator — PATH
Locations (2):
- Kenya (2):
  - Kisumu District Hospital, Kisumu, Nyanza
  - New Nyanza Provincial General Hospital, Kisumu, Nyanza

REFERENCES:
- See also: Related Info — http://www.mbiodx.com/technology/